CLINICAL TRIAL: NCT03083652
Title: Effects of Neuromuscular Electrical Stimulation on Exercise Capacity in Respiratory Critically Ill Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Joan-Daniel Martí Romeu, Principal Investigator, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: UVIR
Record Dates: First submitted 2017-02-28; First posted 2017-03-20 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Critical Illness Myopathy
Keywords: physiotherapy; neuromuscular electrical stimulation; exercise capacity
MeSH Terms: interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Sham Comparator): Conventional physiotherapy with NMEs device not activated
  Interventions: Other: Sham
- Intervention (Experimental): Conventional physiotherapy with daily 30-minutes NMEs (5 days/week)
  Interventions: Device: Neuromuscular electrical stimulation

INTERVENTIONS:
Device: Neuromuscular electrical stimulation — Neuromuscular electrical stimulation (30 minutes per day, 5 days/week) of the quadriceps femoris and gluteus maximus
  Arms: Intervention
Other: Sham — Conventional physiotherapy with NMES device NOT activated
  Arms: Control

SUMMARY:
Neuromuscular electrical stimulation (NMES) implemented during the intensive care unit(ICU) stay may improve exercise capacity and prevent muscular weakness in critically ill patients with respiratory disease. Main objective: To evaluate, in respiratory critically ill patients, the effects of a conventional physiotherapy program with or without additional NMES applied only during the ICU stay on exercise capacity. Design: Randomized, controlled, double-blind clinical trial on patients (>18yo) with diagnosis on admission of acute or acute on chronic respiratory disease, on mechanical ventilation (MV) > 72h and expected MV > 24h. Intervention: Conventional physiotherapy with or without 30-minutes (5days/week) on quadriceps femoris and gluteus maximus. Patients in the control group will follow the same protocol but the device will not be activated. Measures: Demographic data, body composition through bioelectrical impedance analysis (BIA), and functional capacity before admission through Barthel scale will be registered upon inclusion. Exercise capacity through test sit-to stand, muscular strength through Medical Research Council (MRC) score and dynamometry, body composition through BIA, and functional capacity through Barthel scale will be obtained at ICU and hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis at admission: acute or acute on chronic respiratory disease
* Mechanical ventilation > 72h at inclusion
* Expected mechanical ventilation > 24h
* Informed consent

Exclusion Criteria:

* Patients re-admitted to ICU (no hospital discharge)
* Exitus or transfer to another service/hospital
* Respiratory instability [Inspired fraction of oxygen (FIO2) >60% or positive end-expiratory pressure (PEEP) >10 cmH2O] and/or hemodynamic instability [Mean arterial pressure ( MAP)<60mmHg although vasoactive drugs] during > 24h.
* Pregnancy
* Neuromuscular disease before admission
* Skin lesions
* Limitation of therapeutic effort
* Mental and/or physical limitation to understand/realize tests for evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-02-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Exercise capacity | <48h from ICU discharge
  Test sit-to-stand
Exercise capacity | 24h before hospital discharge
  Test sit-to-stand

SECONDARY OUTCOMES:
Muscle strength | 1st day in which collaboration of the patient is ensured (through standardized 5 questions)
  MRC score
Muscle strength | <48 from ICU discharge
  MRC score
Muscle strength | 24h before hospital discharge
  MRC score
Muscle strength | 1st day in which collaboration of the patient is ensured (through standardized 5 questions)
  Dynamometry
Muscle strength | <48 from ICU discharge
  MRC score and dynamometry
Muscle strength | 24h before hospital discharge
  MRC score and dynamometry
Body composition (fat free mass) | <48h from inclusion
  Bioelectrical impedance
Body composition (fat free mass) | <48 from ICU discharge
  Bioelectrical impedance
Body composition (fat free mass) | 24h before hospital discharge
  Bioelectrical impedance
Functional Capacity | <24h from inclusion
  Barthel scale
Functional Capacity | 24h before hospital discharge
  Barthel scale

CONTACTS AND LOCATIONS:
Overall Officials: Joan-Daniel Martí, Pt,PhD, Principal Investigator — Physiotherapist
Locations (1):
- Unidad de Vigilancia Intensiva Respiratoria (UVIR), Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Abdellaoui A, Prefaut C, Gouzi F, Couillard A, Coisy-Quivy M, Hugon G, Molinari N, Lafontaine T, Jonquet O, Laoudj-Chenivesse D, Hayot M. Skeletal muscle effects of electrostimulation after COPD exacerbation: a pilot study. Eur Respir J. 2011 Oct;38(4):781-8. doi: 10.1183/09031936.00167110. Epub 2011 Feb 24. PMID 21349913
- [Result] Zanotti E, Felicetti G, Maini M, Fracchia C. Peripheral muscle strength training in bed-bound patients with COPD receiving mechanical ventilation: effect of electrical stimulation. Chest. 2003 Jul;124(1):292-6. doi: 10.1378/chest.124.1.292. PMID 12853536